CLINICAL TRIAL: NCT06029491
Title: The Pivotal Study of RapidPulseTM Aspiration System as Frontline Approach for Patient With Acute Ischemic Stroke Due to Large Vessel Occlusions
Brief Title: The Pivotal Study of RapidPulseTM Aspiration System
Acronym: PIVOTAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RapidPulse, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0002
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; Large Vessel Occlusion; Mechanical Thrombectomy; Neurovascular Intervention
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Thrombectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Arm (Experimental): Each subject will undergo baseline evaluation for acute ischemic stroke due to large vessel occlusion, per standard of care and undergo mechanical thrombectomy procedure, aspiration to remove the thrombus in the neuro-vasculature using the RapidPulseTM Aspiration System.
  Interventions: Device: RapidPulseTM Aspiration System

INTERVENTIONS:
Device: RapidPulseTM Aspiration System — The RapidPulseTM Aspiration System is designed to remove occlusive thrombus from the occluded cerebral vasculature using precisely pulsed aspiration. The system is comprised of the multi-use, non-sterile RapidPulseTM Aspiration Pump, the single use, sterile RapidPulseTM Tube set, the single use, non-sterile RapidPulseTM Collection Canister and the single use, sterile RapidPulseTM 071 Catheter.
  Other Names: Aspiration Thrombectomy; Thrombectomy

SUMMARY:
The goal of this clinical trials is to demonstrate the safety and effectiveness for the RapidPulseTM Aspiration System in patients experiencing acute ischemic stroke within 8 hours of symptom onset or last seen normal. Subjects will undergo mechanical thrombectomy (a procedure to remove a clot in the brain which is preventing blood flow), with the RapidPulseTM Aspiration System. Participation in the trial is for 90 days.

DETAILED DESCRIPTION:
The purpose of this prospective, open label clinical trials is to demonstrate the safety and effectiveness for the RapidPulseTM Aspiration System as frontline approach in the treatment of large vessel occlusions in patients experiencing Acute Ischemic Stroke within 8 hours of symptom onset or last seen normal. The target sample size for this clinical trial is 170 subjects enrolled in up to 30 sites globally. The maximum number of subjects that may be enrolled is 340. Subjects will undergo mechanical thrombectomy procedure and will have postoperative assessments completed at 24 hours and on day 5-7 or hospital discharge (whichever comes first). The final study visit will occur approximately 90 days after the index event. The primary effectiveness endpoint is the proportion of patients who achieve First Pass Reperfusion Effect (FPE) as defined by modified treatment in cerebral infarction score (mTICI) ≥ 2c after the first pass as assessed by an independent Imaging Core Lab. The primary safety endpoint is the proportion of patients with symptomatic ICH (sICH) at 24 hours post-thrombectomy as assessed by a central events committee (CEC).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years
* Clinical diagnosis of acute ischemic stroke with NIH Stroke Scale (NIHSS) score ≥ 6
* Able to be treated within 8 hours of symptom onset or last known normal (LKN)
* Able to be treated within 120 minutes from the time of the qualifying baseline CT/MR image
* Pre-morbid Modified Rankin Scale (mRS) score 0-1
* Angiographic confirmation of large vessel occlusion (LVO) in the anterior (intracranial ICA or MCA M1 or M2 segments) or posterior circulation (vertebral or basilar arteries) as confirmed by digital subtraction angiography (DSA) irrespective of IV thrombolysis administration
* Candidate to receive treatment with ADAPT technique (Direct Aspiration First-Pass Technique)

Exclusion Criteria:

* Intracranial Hemorrhage (ICH)
* Alberta Stroke Program Early CT Score (ASPECTS) <6
* Intracranial Atherosclerotic Disease (ICAD)
* Multiple or tandem occlusions
* Life expectancy less than 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Rate of First Pass Reperfusion Effect (FPE) | Intra-procedural
  The proportion of patients who achieve First Pass Reperfusion Effect (FPE) as defined by mTICI ≥ 2c after the first pass
Rate of symptomatic intracranial hemorrhage (sICH) | Post-procedural (24 hours post-thrombectomy)
  The proportion of patients with symptomatic ICH (sICH) at 24 hours post-thrombectomy

SECONDARY OUTCOMES:
Rate of reperfusion after all study device passes | Intra-procedural
  Proportion of patients who achieve mTICI ≥ 2b within a maximum of 3 passes with Study Device
Modified Rankin Scale (mRS) at 90 days post treatment | Post-procedure (90 days post-thrombectomy)
  Proportion of patients who achieve mRS ≤2 at 90-days post treatment.

OTHER OUTCOMES:
Rate of modified First Pass Reperfusion Effect (mFPE) after one reperfusion attempt | Intra-procedural
  Modified First Pass Reperfusion Effect (mFPE) as defined by mTICI ≥ 2b after one device pass
Final reperfusion effect | Intra-procedural
  Final mTICI ≥ 2b after all passes (including any rescue therapy) at procedure conclusion
Time to reperfusion | Intra-procedural
  Time from arterial puncture (procedure initiation) to achieve mTICI ≥ 2b using first line aspiration treatment.
Rate of major early neurological recovery | Post-procedure (24 hours post-thrombectomy)
  Proportion of patients with major early neurological recovery at 24-hours as defined by reduction in National Institutes of Health Stroke Scale (NIHSS) score from baseline of at least 8 points or reaching NIHSS 0-1.
  *NIHSS ranges from 0 to 42, with higher scores indicating greater neurological deficit.
Incidence of Serious Adverse Events (SAEs) | Intra-procedural to post-procedure (through 90 days post-thrombectomy)
  All device-related and procedure-related serious adverse events
Incidence of all cause mortality | Intra-procedural to post-procedure (through 90 days post-thrombectomy)
  All-cause mortality assessed through 90 days post index procedure.
Incidence of device related vasospasm | Intra-procedural
  Device-related vasospasm
Incidence of embolism in new territory | Intra-procedural
  Embolism in new territory determined based on procedural angiogram
Incidence of all intracranial hemorrhage | Post-procedural (24 hours post-thrombectomy)
  Any intracranial hemorrhage according to the Heidelberg classification at 24-hours

CONTACTS AND LOCATIONS:
Overall Officials: Raul G Nogueira, MD, Principal Investigator — University of Pittsburgh Medical Center Stroke Institute; Marc Ribó, MD, Principal Investigator — Hospital Universitari Vall d' Hebron
Locations (30):
- United States (18):
  - Providence Saint John's Medical Foundation, Torrance, California
  - Yale University, New Haven, Connecticut
  - Baptist Health Research Institute, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University at Grady, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Advocate Aurora Research Institute, Park Ridge, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - State University of Iowa, Iowa City, Iowa
  - Washington University, St Louis, Missouri
  - Cooper Health System, Camden, New Jersey
  - State University of New York at Buffalo, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - UPMC, Pittsburgh, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Semmes Murphey Foundation - Baptist Memorial Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Valley Baptist Medical Center - Harlingen, Harlingen, Texas
- France (3):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
- Spain (8):
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Universitari Vall d' Hebron, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
- Istanbul Aydan Universitesi VM Medical Park Florya Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No